CLINICAL TRIAL: NCT02914483
Title: Women's Heart Attack Research Program: Stress Ancillary Study; Telephone-Based Stress Management for Women With Myocardial Infarction
Brief Title: Women's Heart Attack Research Program: Stress Ancillary Study
Acronym: HARP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-01104-1
Record Dates: First submitted 2016-09-20; First posted 2016-09-26 (Estimated); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; Women; Stress Management
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (EUC) (Other)
  Interventions: Behavioral: Enhanced Usual Care; Diagnostic Test: Actigraph
- Stress Management (Other)
  Interventions: Behavioral: Stress Management; Diagnostic Test: Actigraph

INTERVENTIONS:
Behavioral: Enhanced Usual Care — Participants randomized into the EUC group will complete 8 weekly individual sessions by phone. Each weekly session consists of: brief check-in and review of AHA brochure- "Women, Heart Disease and Stroke".
  Other Names: EUC
  Arms: Enhanced Usual Care (EUC)
Behavioral: Stress Management — Participants randomized into the stress management group will complete 8 weekly group sessions by phone. The intervention is a telephone adaptation of mindfulness-based cognitive therapy (MBCT) and focuses on building cognitive-behavioral and mindfulness skills to help manage and cope with stress. Each hour-long weekly session consists of: check-in, instruction, skill building, discussion, and home-based practice assignment.
  Arms: Stress Management
Diagnostic Test: Actigraph — The Actigraph (wGT3X-BT) will monitor sleep activity and will be worn by participants for 7 days, pre- and post stress based intervention.
  Other Names: 'Sleep Watch'

SUMMARY:
The Women's HARP study is a multi-center study focusing on women with clinical presentation of myocardial infarction (MI). Women will complete stress questionnaires following presentation to the medical center with elevated cardiac enzymes and abnormal electrocardiograms (ECGs). 2 months following MI, participants will be screened for the Stress Ancillary Study and enrolled if an elevated level of perceived stress is reported. After completing baseline assessments, participants will be randomized to Enhanced Usual Care (EUC) or stress management for 8 weeks. Participants will be followed for 6 months.

DETAILED DESCRIPTION:
Women's HARP is a multi-center, observational study which enrolls women with MI who are referred for cardiac catheterization. During the MI hospitalization, questionnaires will be administered to assess psychosocial stress leading up to the event (MI). Participants will also have the option to enroll in the HARP-Stress Ancillary Study and HARP-Platelet Sub-Study. Two months following MI, participants may be screened for the Stress Ancillary Study. Women with elevated perceived stress at screening will be enrolled. Patients will complete baseline assessments (self-report questionnaires and 7 days of wrist actigraphy) and then will be randomized to group-based stress management or to enhanced usual care (EUC). Both study arms involve 8 weekly phone sessions delivered by trained facilitators. Following intervention, participants in both study arms will repeat self-report questionnaires and 7 days of wrist actigraphy. Anticipate enrollment of approximately 200 women to meet target of 144 qualified women.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic symptoms compatible with diagnosis of MI, such as chest pain or anginal equivalent symptoms at rest or new onset exertional anginal equivalent symptoms
* Objective evidence of MI (either or both of the following):

  * Elevation of troponin to above the laboratory upper limit of normal
  * ST segment elevation of ≥1mm on 2 contiguous ECG leads
* Willing to provide informed consent and comply with all aspects of the protocol
* Age ≥ 21 years
* Female sex
* PSS-4 score ≥6 at 2 month follow up visit after MI

Exclusion Criteria:

* Alternate explanation for troponin elevation, such as hypertensive urgency, acute exacerbation of heart failure, chronic elevation due to kidney disease, pulmonary embolism, cardiac trauma.
* Moderately severe or severe depressive symptoms (PHQ-9 ≥ 15)
* Active suicidal ideation (PHQ-9 item #9 or otherwise reported during screening)
* History of or current diagnosis of psychosis (EHR review)
* Significant cognitive impairment (EHR review or evident during screening)
* Current participation in another behavioral clinical trial.

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS-10) scores | 6 months
  6-month change in perceived stress as measured by Perceived Stress Scale (PSS-10)

SECONDARY OUTCOMES:
Short Form (SF-12) Score | 6 months
  6-month change in health-related quality of life as measured by the 12-Item Short Form Health Survey (SF-12)
Seattle Angina Questionnaire-7 Score (SAQ-7) | 6 months
  6-month change in disease-specific health status as measured by the Seattle Angina Questionnaire (SAQ-7)
Patient Health Questionnaire (PHQ-9) | 6 months
  6-month change in depressive symptoms as measured by the Patient Health Questionnaire (PHQ-9)
Sleep quality | 6 months
  6-month change in sleep efficiency as measured by wrist actigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Harmony R Reynolds, MD, Principal Investigator — NYU Langone Medical Center
Locations (14):
- United States (12):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Univeristy of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Dartmouth-Hitchcock, Lebanon, New Hampshire
  - NYU Winthrop, Mineola, New York
  - NYU Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Seton Heart (Ascension) - University of Texas, Austin, Austin, Texas
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - University of Calgary, Calgary

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared after the end of the study.

REFERENCES:
- [Derived] Spruill TM, Reynolds HR, Dickson VV, Shallcross AJ, Visvanathan PD, Park C, Kalinowski J, Zhong H, Berger JS, Hochman JS, Fishman GI, Ogedegbe G. Telephone-based mindfulness training to reduce stress in women with myocardial infarction: Rationale and design of a multicenter randomized controlled trial. Am Heart J. 2018 Aug;202:61-67. doi: 10.1016/j.ahj.2018.03.028. Epub 2018 Apr 21. PMID 29864732